CLINICAL TRIAL: NCT06149026
Title: Comparison of the Effect of Two Interventions on Liver Frailty Index in Pre-frail and Frail Cirrhotic Patients Enlisted for Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Diego Reyes, Fellowship of gastroenterology, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FrailtyRCT
Record Dates: First submitted 2023-08-17; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Cirrhosis, Liver
Keywords: liver transplant; cirrhosis; nutrition; physical therapy; frailty; quality of life
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis; Frailty | interventions — Restraint, Physical; Nutrition Therapy

STUDY DESIGN:
Intervention Model Description: The goal of this prospective, double blind randomized clinical trial is to compare the effectiveness of two interventions in improve frailty (measured by Liver Frailty Index) and quality of life (measured by Chronic Liver Disease Questionnaire - CLDQ) in listed patients with cirrhosis.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A person who do not participate in the recruitment and the evaluation of the patients randomize a number for each patient. If the number is even, the patient belongs to the intervention group and if the number is odd, the patient belongs to the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group will receive written, detailed, and standardized instructions on nutritional recommendations and physical activity at visit 1. Patients will have follow-up evaluations by a physician to reinforce adherence and make necessary adjustments for compliance with nutritional requirements. Nutritional intake reminder surveys will be conducted during the last 24 hours (E24H) at weeks 0, 4, 8 and 12.
- Intervention group (Experimental): Intervention group consisting of physical therapy guided by a kinesiologist for 10 sessions during which the patient will be trained to maintain physical activity three times a week. In addition, patients will be evaluated by a nutritionist who will give specific indications regarding the quality, quantity, and timing of food intake, as well as the daily frequency of food consumption. Patients will have two follow-ups by a nutritionist (week 4 and 8) to check adherence and make the necessary adjustments to meet nutritional requirements. Nutritional intake reminder surveys will be conducted during the last 24 hours (E24H) at weeks 0, 4, 8 and 12.)
  Interventions: Other: Physical and nutritional therapy

INTERVENTIONS:
Other: Physical and nutritional therapy — The patients will be evaluated and followed by a nutritionist and a physical therapist for 12 weeks. In that time, the patients will receive workouts according to their evaluations and a specific nutritional guide according to the nutritionist's evaluations.
  Arms: Intervention group

SUMMARY:
The goal of this prospective, double blind randomized clinical trial is to compare the effectiveness of two interventions in improve frailty (measured by Liver Frailty Index) and quality of life (measured by Chronic Liver Disease Questionnaire - CLDQ) in listed patients with cirrhosis.

The main questions it aims to answer are:

* if the intervention group (physical and nutritional therapy) could improve LFI over control group (physical and nutritional counseling).
* if the intervention group could improve secondary outcomes as CLDQ, hand grip and gait velocity.

Participants will be evaluated in a registry of basal variables such as demographic factors, weight, height and brachial circumference, comorbidities, MELD and MELD-Na, Child Pugh classification, general blood exams, etiology of cirrhosis, presence of hepatocellular carcinoma, ascites, or hepatic encephalopathy and their basal LFI, gait velocity, hand grip and CLDQ. The participants will be randomized in an intervention group or in a control group at the same time of their first evaluation and will receive the group instructions depending on what group the participants belong, and will be evaluated at 4 weeks, 8 weeks, and 12 weeks with applying LFI, measuring of gait velocity, hand grip and a nutritional survey with the intake in the last 24 hours. Finally, researchers will compare interventional group with control group if the first group could improve frailty, measured by Liver Frailty Index and the secondary outcomes with the nutritional and physical therapy.

DETAILED DESCRIPTION:
Comparison of the effect of two interventions on Liver Frailty Index in pre-frail and frail cirrhotic patients enlisted for liver transplantation.

Frailty is a concept derived from geriatrics that translates a reduction in the physiological reserve of various organs and systems (immune, musculoskeletal, endocrine, neurological, etc.) and a greater vulnerability to stressors. It is present in up to one fifth of cirrhotic patients listed for liver transplantation and its determination has been independently related to adverse outcomes. On the other hand, it is closely linked to the concept of sarcopenia, which translates into a reduction of skeletal muscle mass and function. However, there is a proportion of frail patients who are not sarcopenic (patients with sarcopenia) and not all sarcopenic patients are frail so sarcopenia and frailty are not equivalent concepts, although both are related.

In cirrhosis, the presence of frailty and sarcopenia are conditions that may be determined by a multiplicity of factors such as the presence of hepatic encephalopathy, ascites, poor nutrition, sedentary lifestyle, aging, endocrinological factors, hospitalizations, comorbidities, and also socioeconomic and environmental factors. Sarcopenia could be measured employing several methods. One of the most validated is the determination of the skeletal muscle index, which adjusts the area of skeletal muscle at L3 level by height. Thus, a woman is considered sarcopenic if she has an index lower than 39 cm2/m2 and, in men, when it is lower than 50 cm/m2. This index is related to the patient prognosis. Thus, according to this the survival of sarcopenic patients is always lower when adjusted for other variables, especially in women.

Nevertheless, sarcopenia fails to capture spheres that the concept of frailty consider and that influence the prognosis of patients even in the absence of sarcopenia. There is a multiplicity of instruments that allow to establish the diagnosis of frailty, some very simple and quick to perform, such as the Karnofsky scale (although it has a large subjective component) and others more complex and objective, although demanding in time and resources, such as the cardiopulmonary exercise test (CPET). Other tests evaluated are: Clinical Frailty Scale (CFS), Instrumental Activities of Daily Living (IADL), Fried Frailty Phenotype (FFP), 6 Minute Walk Test (6MWT), Dynamometer Prehension Test (handgrip) or gait speed. The choice of the test to be performed should be based on the simplicity of the test, the need for available instruments, the determination of objective variables, reproducibility, cost, time available and the prognostic significance of the test.

A recent study conducted by our group evaluated the prognostic significance of the presence of frailty assessed by FFP. A total of 126 cirrhotic patients were included, 65.1% of whom were diagnosed as frail. The main etiologies were MAFLD (Metabolic dysfunction-associated fatty liver disease), alcohol liver disease and hepatitis C virus infection. The mean age was 64±8.3 years, 47.6% were women, median MELD-Na 15[12-17] and median follow-up was 881 [349-1,277] days. Interestingly, mortality in frail patients was markedly higher than in robust patients i.e., 26.1% versus 5.9% at 12 months, 47.6% versus 12.0% at 24 months, and 68.2% versus 20.6% at 48 months, respectively (p < 0.001). Additionally, patients with reduced gait speed (less than or equal to 0.8 meters/second) also had higher mortality (32.8% versus 13.3% at 12 months, 58.9% versus 26.2% at 24 months, and 79.9% versus 40.8% at 48 months respectively; p < 0.001). Moreover, multivariate analysis showed that the presence of frailty and low gait speed were related to mortality independent of liver function. Thus, the presence of frailty conferred an increased risk of death with any degree of liver dysfunction.

In the study, FFP was used because it meets the requirements and it had a significant experience in other similar studies. Nonetheless, it would be of greater interest to apply a test specifically designed for patients with chronic liver disease and that adjusts to their peculiarities.

The Liver Frailty Index (LFI) is a test developed to be used specifically in patients with cirrhosis, evaluates objective variables, requires simple instruments, is reproducible, widely available and requires few time to be performed. In addition, it predicts the survival of listed patients. The LFI includes the measurement of prehension strength, a squat test (time required to perform 5 squats) and a balance test with parallel, semi-tandem and tandem feet and provides a score (continuous variable). Thus, when the score is less than 3.2 patients are considered robust, if it is 3.2 to 4.4 the participants are considered pre-fragile and if it is 4.5 or more patients are considered fragile.

Recently, the LFI was used in a randomized controlled trial in cirrhotic patients comparing the use of an exercise program versus standard medical care. Although the trial was negative possibly due to low patient adherence, the use of LFI allowed objective assessment of patient progress and the effect of the intervention without using subjective variables and with a test specifically designed for patients with cirrhosis.

It is interesting to note that current studies have attempt to evaluate the effectiveness of interventions to improve frailty in patients with cirrhosis without discriminating those who are frail or pre-frail from those who are robust. Thus, it is not possible to really know what proportion of the patients included were non-robust and if the interventions are effective in the specific subgroup of patients.

Therefore, a trial was designed to evaluate the effectiveness of an intervention consisting of physical and nutritional therapy compared to physical and nutritional counseling over a 12-week period. Unlike the previously described studies, this study will only enroll pre-fragile and frail patients according to the LFI.

This is a randomized trial which will attempt to evaluate if there is a difference between an intervention that corresponds to our standard behavior but intensified in terms of providing very detailed information and periodic reinforcement and another intervention that will consist of personalized physical training associated with nutritional assistance directed to the specific patient and with periodic consultations.

The potential results of this study will be interesting considering that if any of the interventions is superior it should prefer it, but if both are similar, the most cost effective one should be choose.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of cirrhosis.
2. Over 50 years old.
3. Liver Frailty Index of 3.2 points or more.
4. Ability to follow instructions.
5. Ability to consent to study entry.

Exclusion Criteria:

1. Grade 3 or 4 hepatic encephalopathy.
2. Untreated HIV infection.
3. Previous liver transplant.
4. Inability to walk.
5. Extrahepatic diseases that limit mobility (e.g., neurological or musculoskeletal).
6. Advanced cardiac, renal or pulmonary disease.
7. Expectation of being transplanted during the study period.
8. Hepatocarcinoma (HCC) exceeding the Milan criteria.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Liver Frailty Index | 12 weeks
  The Liver Frailty Index (LFI) is a test developed to be used specifically in patients with cirrhosis, evaluates objective variables, requires simple instruments, is reproducible, widely available and requires few time to be performed. In addition, it predicts the survival of listed patients.

SECONDARY OUTCOMES:
Chronic Liver Disease Questionnaire | 12 weeks
  Test to evaluate the quality of life in cirrhotic patients.
Gait velocity | 12 weeks
  Velocity of the gait of the cirrhotic patients with a walking speed test in four meters
Hand grip | 12 weeks
  Measure of the hand grip with a dynamometer. The prehension strength recorded is the average of 3 prehension attempts with maximal strength.

CONTACTS AND LOCATIONS:
Locations (1):
- Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Yes
The plan will be to share the information of the protocol, the statistical analysis that the investigators will do with the data and the way of measuring the outcomes and the characteristics of the participants with their demographic data and the description of the data related with their comorbidities and cirrhosis. In a supplementary material, the investigators will add the informed consent form.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available when the study will be published in a journal in a supplementary material.
Access Criteria: The access will be defined by the journal.

REFERENCES:
- [Background] Tandon P, Montano-Loza AJ, Lai JC, Dasarathy S, Merli M. Sarcopenia and frailty in decompensated cirrhosis. J Hepatol. 2021 Jul;75 Suppl 1(Suppl 1):S147-S162. doi: 10.1016/j.jhep.2021.01.025. PMID 34039486
- [Background] Puchades Renau L, Herreras Lopez J, Cebria I Iranzo MA, Cezon Serrano N, Di Maira T, Berenguer M. Frailty and Sarcopenia in Acute-on-Chronic Liver Failure. Hepatol Commun. 2021 May 4;5(8):1333-1347. doi: 10.1002/hep4.1722. eCollection 2021 Aug. PMID 34430779
- [Background] Laube R, Wang H, Park L, Heyman JK, Vidot H, Majumdar A, Strasser SI, McCaughan GW, Liu K. Frailty in advanced liver disease. Liver Int. 2018 Dec;38(12):2117-2128. doi: 10.1111/liv.13917. Epub 2018 Jul 15. PMID 29935102
- [Background] Carey EJ, Lai JC, Wang CW, Dasarathy S, Lobach I, Montano-Loza AJ, Dunn MA; Fitness, Life Enhancement, and Exercise in Liver Transplantation Consortium. A multicenter study to define sarcopenia in patients with end-stage liver disease. Liver Transpl. 2017 May;23(5):625-633. doi: 10.1002/lt.24750. PMID 28240805
- [Background] Lai JC, Sonnenday CJ, Tapper EB, Duarte-Rojo A, Dunn MA, Bernal W, Carey EJ, Dasarathy S, Kamath BM, Kappus MR, Montano-Loza AJ, Nagai S, Tandon P. Frailty in liver transplantation: An expert opinion statement from the American Society of Transplantation Liver and Intestinal Community of Practice. Am J Transplant. 2019 Jul;19(7):1896-1906. doi: 10.1111/ajt.15392. Epub 2019 May 8. PMID 30980701
- [Background] Ney M, Haykowsky MJ, Vandermeer B, Shah A, Ow M, Tandon P. Systematic review: pre- and post-operative prognostic value of cardiopulmonary exercise testing in liver transplant candidates. Aliment Pharmacol Ther. 2016 Oct;44(8):796-806. doi: 10.1111/apt.13771. Epub 2016 Aug 19. PMID 27539029
- [Background] Soto R, Diaz LA, Rivas V, Fuentes-Lopez E, Zalaquett M, Bruera MJ, Gonzalez C, Mezzano G, Benitez C. Frailty and reduced gait speed are independently related to mortality of cirrhotic patients in long-term follow-up. Ann Hepatol. 2021 Nov-Dec;25:100327. doi: 10.1016/j.aohep.2021.100327. Epub 2021 Feb 14. PMID 33596465
- [Background] Lai JC, Covinsky KE, Dodge JL, Boscardin WJ, Segev DL, Roberts JP, Feng S. Development of a novel frailty index to predict mortality in patients with end-stage liver disease. Hepatology. 2017 Aug;66(2):564-574. doi: 10.1002/hep.29219. Epub 2017 Jun 28. PMID 28422306
- [Background] Williams FR, Berzigotti A, Lord JM, Lai JC, Armstrong MJ. Review article: impact of exercise on physical frailty in patients with chronic liver disease. Aliment Pharmacol Ther. 2019 Nov;50(9):988-1000. doi: 10.1111/apt.15491. Epub 2019 Sep 9. PMID 31502264
- [Background] Haugen CE, McAdams-DeMarco M, Verna EC, Rahimi RS, Kappus MR, Dunn MA, Volk ML, Gurakar A, Duarte-Rojo A, Ganger DR, O'Leary JG, Ladner D, Garonzik-Wang J, Segev DL, Lai JC. Association Between Liver Transplant Wait-list Mortality and Frailty Based on Body Mass Index. JAMA Surg. 2019 Dec 1;154(12):1103-1109. doi: 10.1001/jamasurg.2019.2845. PMID 31509169
- [Background] Lai JC, Dodge JL, Kappus MR, Wong R, Mohamad Y, Segev DL, McAdams-DeMarco M. A Multicenter Pilot Randomized Clinical Trial of a Home-Based Exercise Program for Patients With Cirrhosis: The Strength Training Intervention (STRIVE). Am J Gastroenterol. 2021 Apr;116(4):717-722. doi: 10.14309/ajg.0000000000001113. PMID 33982941
- [Background] Hughes MJ, Hackney RJ, Lamb PJ, Wigmore SJ, Christopher Deans DA, Skipworth RJE. Prehabilitation Before Major Abdominal Surgery: A Systematic Review and Meta-analysis. World J Surg. 2019 Jul;43(7):1661-1668. doi: 10.1007/s00268-019-04950-y. PMID 30788536
- [Background] Zenith L, Meena N, Ramadi A, Yavari M, Harvey A, Carbonneau M, Ma M, Abraldes JG, Paterson I, Haykowsky MJ, Tandon P. Eight weeks of exercise training increases aerobic capacity and muscle mass and reduces fatigue in patients with cirrhosis. Clin Gastroenterol Hepatol. 2014 Nov;12(11):1920-6.e2. doi: 10.1016/j.cgh.2014.04.016. Epub 2014 Apr 24. PMID 24768811
- [Background] Williams FR, Vallance A, Faulkner T, Towey J, Durman S, Kyte D, Elsharkawy AM, Perera T, Holt A, Ferguson J, Lord JM, Armstrong MJ. Home-Based Exercise in Patients Awaiting Liver Transplantation: A Feasibility Study. Liver Transpl. 2019 Jul;25(7):995-1006. doi: 10.1002/lt.25442. Epub 2019 Jun 6. PMID 30859755
- [Background] Chen HW, Ferrando A, White MG, Dennis RA, Xie J, Pauly M, Park S, Bartter T, Dunn MA, Ruiz-Margain A, Kim WR, Duarte-Rojo A. Home-Based Physical Activity and Diet Intervention to Improve Physical Function in Advanced Liver Disease: A Randomized Pilot Trial. Dig Dis Sci. 2020 Nov;65(11):3350-3359. doi: 10.1007/s10620-019-06034-2. Epub 2020 Jan 6. PMID 31907774
- [Background] Ng TP, Feng L, Nyunt MS, Feng L, Niti M, Tan BY, Chan G, Khoo SA, Chan SM, Yap P, Yap KB. Nutritional, Physical, Cognitive, and Combination Interventions and Frailty Reversal Among Older Adults: A Randomized Controlled Trial. Am J Med. 2015 Nov;128(11):1225-1236.e1. doi: 10.1016/j.amjmed.2015.06.017. Epub 2015 Jul 6. PMID 26159634
- [Background] Roman E, Garcia-Galceran C, Torrades T, Herrera S, Marin A, Donate M, Alvarado-Tapias E, Malouf J, Nacher L, Serra-Grima R, Guarner C, Cordoba J, Soriano G. Effects of an Exercise Programme on Functional Capacity, Body Composition and Risk of Falls in Patients with Cirrhosis: A Randomized Clinical Trial. PLoS One. 2016 Mar 24;11(3):e0151652. doi: 10.1371/journal.pone.0151652. eCollection 2016. PMID 27011355
- [Background] Kruger C, McNeely ML, Bailey RJ, Yavari M, Abraldes JG, Carbonneau M, Newnham K, DenHeyer V, Ma M, Thompson R, Paterson I, Haykowsky MJ, Tandon P. Home Exercise Training Improves Exercise Capacity in Cirrhosis Patients: Role of Exercise Adherence. Sci Rep. 2018 Jan 8;8(1):99. doi: 10.1038/s41598-017-18320-y. PMID 29311671
- [Background] Lattanzi B, Bruni A, Di Cola S, Molfino A, De Santis A, Muscaritoli M, Merli M. The Effects of 12-Week Beta-Hydroxy-Beta-Methylbutyrate Supplementation in Patients with Liver Cirrhosis: Results from a Randomized Controlled Single-Blind Pilot Study. Nutrients. 2021 Jul 2;13(7):2296. doi: 10.3390/nu13072296. PMID 34371806